CLINICAL TRIAL: NCT01613183
Title: Exploratory Study of Effective Core Formula of Chinese Medicine to Treat Primary Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liyun He, Director, Principal Investigator, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PJZX-001; 81072920 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2012-05-16; First posted 2012-06-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chinese Medicine group (Experimental): Chinese Medicine prescription of one of three prestigious Chinese medicine clinicians
  Interventions: Drug: Chinese herbal Medicine
- placebo group (Placebo Comparator)
  Interventions: Other: the dummy of a Chinese Medicine prescription

INTERVENTIONS:
Drug: Chinese herbal Medicine — The intervention of Chinese Medicine group is not fixed. The clinicians provide the prescription to patient base their own Chinese Medicine theory. Chinese clinicians can adjust the medicinal in prescription based on the condition of patient during the treatment procedure. The prescription of Chinese clinicians' are pure Chinese herb.
  Arms: Chinese Medicine group
Other: the dummy of a Chinese Medicine prescription — Patients in placebo group will receive the dummy of the core drug patterns screened in previous retrospective study. The previous core drug patterns include Fried semen Ziziphi Spinosae, Tuckahoe, Preparation of Polygala, Chinese Angelica root, Lotus heart, White peony root, dried tangerine peel, acorus calamus, Coptis chinensis, and Licorice health.
  Arms: placebo group

SUMMARY:
The objective of this study is to screen the effective core formulation in insomnia treatment with Chinese medicine with a double-blind, randomized, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 65 years,
* meeting the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) of insomnia,
* Spiegel scale score is ≥ 18,
* The informed consent must be obtained from patient

Exclusion Criteria:

* total sleep time ≤ 2 hours,
* secondary insomnia,
* Self-rating Anxiety Scale (SAS) score ≥ 18,
* Beck Depression Inventory (BDI) score ≥ 6,
* having hypertension, diabetes, stroke, and coronary heart disease,
* have drug abuse history,
* pregnancy or preparing to pregnancy,
* used immunotherapy or hormone therapy in past 1 years,
* participating in another clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2
Dates: Start 2012-05

PRIMARY OUTCOMES:
change from baseline in Total Sleep Time (TST) at 4 weeks | baseline and 4 weeks

SECONDARY OUTCOMES:
change from baseline in sleep onset latency at 4 weeks | baseline and 4 weeks
change from baseline in wake time after sleep onset at 4 weeks | baseline and 4 weeks
change from baseline in sleep efficiency at 4 weeks | baseline and 4 weeks
change from baseline in Pittsburgh sleep quality index (PSQI) at 4 weeks | baseline and 4 weeks
change from baseline in Chinese Medicine symptoms and signs at 4 weeks | baseline and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Liyun He, Doctor, Study Chair — China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen hospital, China Academy of Chinese Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Xiong ZY, Lu Y, He LY, Zhang RS, Zhou XZ, Li P, Liu YJ, Zhu JG, Yan SY, Liu BY. Efficacy of Chinese Medicine Treatment Based on Syndrome Differentiation for Primary Insomnia: A Randomized Placebo Controlled Triple-Blinded Trial. Chin J Integr Med. 2024 Oct;30(10):867-876. doi: 10.1007/s11655-024-3661-4. Epub 2024 May 16. PMID 38753273
- [Derived] Yan S, Zhang R, Zhou X, Li P, He L, Liu B. Exploring effective core drug patterns in primary insomnia treatment with Chinese herbal medicine: study protocol for a randomized controlled trial. Trials. 2013 Feb 28;14:61. doi: 10.1186/1745-6215-14-61. PMID 23448313